CLINICAL TRIAL: NCT01263626
Title: Monitoring Cough Device - Step 1 and 2
Brief Title: Cough Monitoring Study
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Medical Director, Vanderbilt University
Other Study IDs: MCD 1-2
Record Dates: First submitted 2010-12-16; First posted 2010-12-21 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Cough; Reflux
Keywords: Cough; Chronic Cough; Reflux
MeSH Terms: conditions — Cough; Gastroesophageal Reflux; Chronic Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cough as Primary Complaint: 1. Male and female volunteers 18 years of age and older
  2. Cough as chief complaint
  3. Referred to the GI clinic to evaluate if reflux is the cause of their chief complaint
  4. pH testing for standard of care purposes
- Healthy Volunteers: 1. Male and female volunteers 18 years of age and older
  2. No history of chronic or acute cough and throat clearing
  3. Ability to read a 5th grade script written in English for approximately 20 minutes

SUMMARY:
The aim of the study is to establish the accuracy of a new device designed specifically to record and detect cough episodes.

Cough is an important defense mechanism of the respiratory tract. The presence of chronic cough may indicate the presence of underlying diseases, including reflux. Despite the increased number of patients suffering from cough in the ENT and GI practice, to date, there has been no method/device to objectively assess the frequency of cough episodes in a given patient.

PULMOTRACK-CC, manufactured by KarmelSonix (Haifa, Israel), has recently introduced an innovative device that is able to record cough episodes and then automatically detect and count them with the help of a specific software program. This study will assess the accuracy of this novel cough monitoring and counting technology and validate potential clinical use in patients with chronic cough.

ELIGIBILITY:
Inclusion Criteria:

Arm 1: healthy volunteers:

1. Male and female volunteers 18 years of age and older
2. No history of chronic or acute cough and throat clearing
3. Ability to read a 5th grade script written in English for approximately 20 minutes

Arm 2: patients:

1. Male and female volunteers 18 years of age and older
2. Cough as chief complaint
3. Referred to the GI clinic to evaluate if reflux is the cause of their chief complaint
4. pH testing for standard of care purposes

Exclusion Criteria:

* Subjects who are not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present to the ENT or GI clinics at Vanderbilt Medical Center with a chief complaint of chronic cough will be eligible for participation in this study. Patients who meet eligibility requirements will be able to participate regardless of sex, social status, or ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of Cough Device | 24 hours post device placement
  The aim of the study is to establish the accuracy of a new device designed specifically to record and detect cough episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaezi, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Francis DO, Slaughter JC, Ates F, Higginbotham T, Stevens KL, Garrett CG, Vaezi MF. Airway Hypersensitivity, Reflux, and Phonation Contribute to Chronic Cough. Clin Gastroenterol Hepatol. 2016 Mar;14(3):378-84. doi: 10.1016/j.cgh.2015.10.009. Epub 2015 Oct 19. PMID 26492842